CLINICAL TRIAL: NCT02311504
Title: OCT Screening of Diabetes Patients: Health Care Research in Secondary Diabetes Care Centers
Brief Title: Eye Screening in German Secondary Diabetes Care Centers
Acronym: DiabCheckophta
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: DCophtaOCTplus14_C
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DiabCheck ophta OCTplus: persons with diabetes undergoing OCT examination
  Interventions: Device: OCT examination

INTERVENTIONS:
Device: OCT examination

SUMMARY:
In patients with confirmed diagnosis of diabetes, an eye examination and a comprehensive survey are conducted after recruitment in secondary diabetes care centers. All patients undergo a comprehensive eye examination including wide-angle fundus photograph and ocular cohaerence tomography. A questionnaire assesses the characteristics (history: diabetes duration, type of treatment), knowledge and personal attitudes of the persons affected. The relevant lab findings were collected from the electronic files.

Main focus of the study is the concordance to the national screening recommendations (last eye exam, presence of retinopathy).

ELIGIBILITY:
Inclusion Criteria:

- diabetes

Exclusion Criteria:

* mental handicap
* in the case of blindness absence of a caregiver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with diabetes in secondary care diabetes centers
Sampling Method: Non-Probability Sample
Enrollment: 831 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
presence of diabetic retinopathy | day

CONTACTS AND LOCATIONS:
Locations (1):
- University Eye Hospital, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Marahrens L, Ziemssen F, Fritsche A, Ziemssen T, Kern R, Martus P, Roeck D. Limited Time from the Diabetes Patients' Perspective: Need for Conversation with the Eye Specialist. Ophthalmologica. 2016;236(3):154-158. doi: 10.1159/000450708. Epub 2016 Oct 5. PMID 27701169